CLINICAL TRIAL: NCT03208751
Title: A 6-months Lifestyle Intervention With Interval and Resistance Exercise in Patients With Coronary Artery Disease and Diabetes Mellitus in a Community Based Setting
Brief Title: Sport as Therapy: a 6-months Lifestyle-Intervention for Patients With Coronary Artery Disease and/or Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Technical University of Munich (Other)
Responsible Party: Principal Investigator, Jeffrey W Christle, Principal investigator, Technical University of Munich
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 5132/11
Record Dates: First submitted 2017-05-26; First posted 2017-07-06 (Actual); Last update posted 2019-07-19 (Actual); Status verified 2019-07

CONDITIONS: Exercise Training; Coronary Artery Disease; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Coronary Artery Disease; Diabetes Mellitus, Type 2 | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: A single-arm intervention with exercise training as secondary prevention strategy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise training (Other): All patients were included in the exercise training group
  Interventions: Behavioral: Exercise training

INTERVENTIONS:
Behavioral: Exercise training — Exercise intervention was divided into 3 phases:
  Phase 1: 6 weeks of moderate continuous training (MCT) 20 to 40 minutes at intensity of 60% of VO2peak, 3 times/week Phase 2: 6 weeks of moderate intensity interval training (MIIT) 30-40 min, intensity 60 to 80% of VO2peak, twice weekly plus at least once weekly MCT home based training Phase 3 (after performing new exercise testing to adapt training intensities): 12 weeks of MIIT 40 min once/week, intensity 60-80/85% of VO2peak, plus at least twice weekly home based MCT. From phase 2, supervised sessions included resistance training of at least 3 muscle groups, 3x15 repetitions at moderate intensity (Borg 12-14).
  Nutritional counseling is offered up to 4 times in 6 months on an individual basis.

SUMMARY:
Regular exercise training has shown to improve exercise capacity in patients with cardiovascular disease. The feasibility and transferability of exercise training in a community based cardiovascular rehabilitation setting is currently less well investigated. The objective of this study is to translate regular exercise training into a community based setting. A 6 months training intervention program with lifestyle counseling is performed, with both supervised training in rehabilitation centres as well as home based training. The aim of the project is to implement this program for a wider patient population and to improve exercise capacity, diastolic function as well as cardiometabolic parameters.

DETAILED DESCRIPTION:
From 2011, patients insured at "Techniker" health insurance company with diagnosed coronary heart disease, heart failure and/or diabetes mellitus are being included in a 6-months training program. Training is performed 3 times weekly for 6 weeks, then twice weekly for another 6 weeks, while patients are asked to do home based training. The last phase of 12 weeks, supervised training is only once/week. Patients are asked to perform exercise training 3-5 times weekly. At the beginning as well as after 3 and 6 months, patients present for medical check-up with cardiorespiratory exercise testing from which training instructions are drawn. Training-intensity begins with moderate continuous training and switches to higher intensity interval training after 6 weeks. Resistance training starts after 6 weeks and is performed within the supervised training. All patients were offered an individual nutritional counseling.

ELIGIBILITY:
Inclusion Criteria:

* Coronary artery disease and/or diabetes mellitus
* Heart failure

Exclusion Criteria:

* all conditions which are not compatible with exercise training:
* severe orthopedic disorders
* severe psychiatric disease
* severe valve insufficiency
* presence of myocardial ischemia (decision made by cardiologist)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2011-04-01 (Actual); Primary Completion 2019-08-01 (Estimated); Study Completion 2020-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in VO2peak in ml/kg/min | 6 months
  Exercise capacity measured by cardiorespiratory exercise testing from start to the end of 6 months training intervention

SECONDARY OUTCOMES:
Change in HbA1c for patients with diabetes | 6 months
  Glycated hemoglobin >5,7 corresponds to glucose intolerance, > 6,5 is diagnosed diabetes mellitus
Change in hsCRP | 6 months
  high sensitivity C-reactive protein, as an inflammation marker and risk marker for further CAD events
Change in E/e' | 6 months
  E/e' is an echocardiographic marker for diastolic function, an E/e' < 8 is considered as normal
Change in quality of life measured by SF-36 | 6 months
  The short form (SF-36) is a validated questionnaire for quality of life, the physical and psychical sum scale are measured
Change in insulin IU | 6 months
  Insulin dosage is measured in IE (international units)
Change in HDL- and LDL- cholesterol as well as triglycerides | 6 months
  all measured in mg/dl
Change in Adiponectin | 6 months
  Adiponectin is an adipokine which is released by fat tissue
Change in Watts at anaerobic threshold VAT | 6 months
  VAT= ventilatory anaerobic threshold, measured by cardiopulmonary exercise testing
Change in Watts at anaerobic threshold RCP | 6 months
  RCP= respiratory compensation point, measured by cardiopulmonary exercise testing
Change in max. Watts | 6 months
  On bicycle ergometry, Watts are measured
Change in max. Watts/kg bodyweight | 6 months
  max. Watts indexed b body weight

CONTACTS AND LOCATIONS:
Overall Officials: Martin Halle, Prof., Study Director — Technical University Munic
Locations (1):
- Klinikum rechts der Isar/ Technische Universitaet Muenchen, Munich, Germany

IPD SHARING:
Plan to Share IPD: No